CLINICAL TRIAL: NCT02914223
Title: Single-center, Open-label Study With 14C-radiolabeled Cenerimod to Investigate the Mass Balance, Pharmacokinetics, and Metabolism Following Single Oral Administration to Healthy Male Subjects
Brief Title: A Study to Evaluate Cenerimod in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AC-064-103
Record Dates: First submitted 2016-09-13; First posted 2016-09-26 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — cenerimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Treatment and observation period (Experimental): On Day 1, subjects will receive a single oral dose of 2 mg 14C-radiolabeled cenerimod. Subjects will be followed for 21 days during which blood, urine, feces, and expired air samples will be collected
  Interventions: Drug: Cenerimod
- Extended observation period (Experimental): In case, radioactivity recovery does not meet the stopping criteria described in the protocol, the subjects will have to come for a maximum of 7 24-h in-clinic visits during which blood, urine, feces, and expired air samples will be collected
  Interventions: Drug: Cenerimod

INTERVENTIONS:
Drug: Cenerimod — Oral formulation of cenerimod (2mg) containing 100 μCi (3.7 MBq) of 14C-radiolabeled cenerimod

SUMMARY:
The main objective of the study is to investigate the rate and routes of elimination of cenerimod and the mass balance in urine, feces, and expired air

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure
* Healthy male subjects aged between 45 and 65 years (inclusive) at screening
* No clinically significant findings on the physical examination at screening
* Body mass index (BMI) of 18.0 to 30.0 kg/m2 (inclusive) at screening
* Systolic blood pressure (SBP) 100-145 mmHg and diastolic blood pressure (DBP) 50-90 mmHg, measured on either arm, after 5 min in the supine position at screening and at Day 1 pre-dose
* Heart rate (HR) 55-90 bpm (inclusive) measured with 12-lead ECG after 5 min in the supine position at screening and at Day 1 pre-dose

Exclusion Criteria:

* Known hypersensitivity to cenerimod or to S1P receptor modulators, or to any excipients of the cenerimod drug formulation
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism, or excretion of the study treatment (appendectomy and herniotomy allowed, cholecystectomy not allowed)
* History or clinical evidence suggestive of active or latent tuberculosis including a positive QuantiFERON®-TB test at screening
* Any cardiac condition or illness (including 12-lead ECG abnormalities) with a potential to increase the cardiac risk of the subject based on the standard 12-lead ECG at screening and at Day 1 pre-dose
* Participation in another study with a radiation burden of > 0.1 mSv and ≤ 1 mSv in the period of 1 year prior to screening; a radiation burden of ≥ 1.1 mSv and ≤ 2 mSv in the period of 2 years prior to screening, etc. (add 1 year per 1 mSv)
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol
* Any immunosuppressive treatment within 6 weeks or within 5 elimination half-lives of the immunosuppressive treatment, whichever is longer, before study treatment administration

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09-01; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Cumulative excretion calculated by summing up the daily radioactivity excretion measured by means of liquid scintillation counting in urine, feces, and expired air (if applicable) | From baseline up to a maximum of 99 days

SECONDARY OUTCOMES:
Cmax (maximum plasma concentration) of 14C-radioactivity in whole blood and plasma | From baseline up to a maximum of 99 days
  Cmax is derived from the observed plasma concentration-time curves
tmax (time to reach Cmax) of 14C-radioactivity in whole blood and plasma | From baseline up to a maximum of 99 days
  Tmax is derived from the observed plasma concentration-time curves
t1/2 (terminal half-life) | From baseline up to a maximum of 99 days
Area under the plasma concentration-time curve (AUC) of 14C-radioactivity in whole blood and plasma | From baseline up to a maximum of 99 days
  AUC is defined for the time intervals from zero to time t of the last measured concentration above the limit of quantification and from zero to infinity
Incidence of safety events of interest | From baseline up to a maximum of 99 days
  Events of interest are any abnormalities in ECG, vital signs or laboratory test results
Number of participants with adverse events (AEs) | From baseline up to a maximum of 99 days
  Treatment-emergent AEs and treatment emergent serious AEs
Cenerimod metabolites profiling in plasma | From baseline up to a maximum of 99 days
  Relative abundance expressed as percent of cenerimod
Cenerimod metabolites profiling in urine | From baseline up to a maximum of 99 days
  Relative abundance expressed as percent of cenerimod
Cenerimod metabolites profiling in feces | From baseline up to a maximum of 99 days
  Relative abundance expressed as percent of cenerimod

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (1):
- PRA Health Science, Groningen, Netherlands